CLINICAL TRIAL: NCT02585830
Title: Investigating the Relationship Between Circadian Phase and Insulin Resistance in Obese Adolescents
Brief Title: Sleep Timing and Insulin Resistance in Adolescents With Obesity
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-0739; UL1TR001082 (NIH)
Record Dates: First submitted 2015-10-22; First posted 2015-10-23 (Estimated); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study examines the relationship between sleep timing and insulin resistance in adolescents with obesity. The investigators also aim to develop a physiologically-based mathematical model of adolescent sleep/wake and circadian interactions.

ELIGIBILITY:
Inclusion Criteria:

* High school students between the ages of 15-19
* BMI > 90th percentile
* Tanner stage 2 or greater

Exclusion Criteria:

* Any medications that affect insulin resistance or sleep (e.g., metformin, hormonal contraception, stimulants, atypical antipsychotics)
* Regular use of melatonin or sleep aids
* A prior diagnosis of obstructive sleep apnea, diabetes (HbA1c > 6.5), liver disease other than non-alcoholic fatty liver disease, pregnancy or breastfeeding
* IQ < 70 or severe mental illness that may impact sleep (e.g., schizophrenia, psychotic episodes)
* Not enrolled in a traditional high school academic program (e.g., home school students)
* Night shift employment
* Travel across more than 2 time zones in the month prior to the study

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents with obesity
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey L Simon, PhD, Principal Investigator — University of Colorado Denver & Children's Hospital Colorado
Locations (1):
- University of Colorado Anschutz Medical Campus/Children's Hospital Colorado, Aurora, Colorado, United States

REFERENCES:
- [Derived] Simon SL, McWhirter L, Diniz Behn C, Bubar KM, Kaar JL, Pyle L, Rahat H, Garcia-Reyes Y, Carreau AM, Wright KP, Nadeau KJ, Cree-Green M. Morning Circadian Misalignment Is Associated With Insulin Resistance in Girls With Obesity and Polycystic Ovarian Syndrome. J Clin Endocrinol Metab. 2019 Aug 1;104(8):3525-3534. doi: 10.1210/jc.2018-02385. PMID 30888398

RESULTS

PARTICIPANT FLOW:
Groups:
- Adolescent Sleep Observation: Home and in-lab observation of sleep and insulin sensitivity
Period: Overall Study
Arm/Group | Adolescent Sleep Observation
Started | 25
Completed | 22
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- Observation: Home and in-lab observation
Arm/Group | Observation
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.48 (1.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 12
  More than one race | 6
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 25
BMI [Mean (Standard Deviation); unit: percentile] — Population: missing data N =4
  percentile
    number analyzed (Participants) | 21
    (all) | 97.04 (2.39)

OUTCOME MEASURES:

1. Primary Outcome: Dim Light Melatonin Onset and Offset
Description: ~1mL saliva was collected at 30- to 60- minute intervals in dim light (<5 lux in the angle of gaze, approximately the light level of candlelight or civil twilight) from approximately 5pm until noon the next day. Dim light melatonin onset (DLMOn) was defined as the linear interpolated clock time at which evening salivary melatonin concentrations increased and remained above a threshold of 3pg/mL. Melatonin offset (DLMOff) was the linear interpolated clock time at which salivary melatonin concentrations fell below this threshold. Later DLMOn and DLMOff are indicative of a later circadian rhythm.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: decimal hours
Arm/Group | Observation
Number analyzed (Participants) | 22
decimal hours
  Dim Light Melatonin Onset | 21.33 (1.47)
  Dim Light Melatonin Offset | 8.32 (1.09)

2. Primary Outcome: Insulin Sensitivity
Description: After an overnight fast, participants completed an oral glucose tolerance test (OGTT) in the morning. Participants consumed a 75g dextrose drink and serum for glucose and insulin concentrations were collected at baseline and every 30 minutes for 3 hours. The homeostatic model assessment for insulin resistance (HOMA-IR) was calculated as [fasting insulin (μU/ml) x fasting glucose (mmol/l)] / 22.5); lower HOMA-IR indicates better insulin sensitivity. The Matsuda Index was calculated as √10,000 / [[fasting insulin (μU/ml) x fasting glucose (mmol/l)] x [mean OSTT insulin (μU/ml) x mean OSTT glucose (mmol/l)]]; high Matsuda Index indicates better insulin sensitivity.
Time Frame: 3 hours
Population: 1 participant with missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Observation
Number analyzed (Participants) | 21
units on a scale
  Homeostatic Model Assessment (HOMA-IR) | 2.9 (2.01)
  Matsuda Index | 4.93 (2.75)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Observation
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT02585830/Prot_SAP_000.pdf